CLINICAL TRIAL: NCT06474637
Title: Prospective Clinical Evaluation of the AEON Endoscopic Stapler Powered Handle and Reload in Primary Sleeve Gastrectomy
Brief Title: Powered Handle Primary Sleeve Gastrectomy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lexington Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endostapler05
Record Dates: First submitted 2024-06-20; First posted 2024-06-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sleeve Gastrectomy
Keywords: LSG (Laparoscopic Sleeve Gastrectomy)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Device: AEON Endoscopic Powered Stapler Handle and Reload

INTERVENTIONS:
Device: AEON Endoscopic Powered Stapler Handle and Reload — The AEON™ Endoscopic Stapler places two triple-staggered rows of titanium staples while simultaneously transecting between the two triple-staggered rows of staples. The size of the staples and staple line length are based on the selection of the Stapler Reload (2.0mm, 2.5mm, 3.25mm, 4.0mm, 5.0mm and 5.5mm).

SUMMARY:
The objective of this prospective, single arm, single-center study is to evaluate patients who are undergoing primary sleeve gastrectomy procedures and are surgically treated with the AEON Endoscopic Powered Handle Stapler and Stapler Reload. The primary endpoint is to assess the percentage of patients who encountered post-operative staple line complications (bleeding or leak), defined as requiring blood transfusion or revision surgery due to staple line complications.

ELIGIBILITY:
Inclusion Criteria:

1. Be within the range of 18-65 years of age
2. Patients undergoing primary sleeve gastrectomy procedures
3. Psychosocially, mentally, and physically able to comply with protocol, post-operative management and follow-up schedule.

Exclusion Criteria:

1. Prior bariatric surgery procedure
2. Sleeve gastrectomy procedure that is planned to be performed via open approach
3. Patients receiving anticoagulant medication(s)
4. Severe heart disease or lung problems
5. Known sensitivity to implant materials
6. Evidence of active (systemic or localized) infection at time of surgery
7. Women who are pregnant or planning to get pregnant in the next 12 months
8. Recent history of known alcohol and/or narcotic abuse
9. Investigational drug or device use within 30 days
10. Any other factors that may contribute, based on professional judgement of the treating surgeon, to the subject being a poor candidate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Post Operative Staple Line Complications | 1 week
  The primary measure of effectiveness and safety will be determined by the incidence of post-operative staple line complications defined as requiring blood transfusion and revision surgery to treat staple line complications.

SECONDARY OUTCOMES:
Hospital Stay | 1 week
  Average hospital stay will be measure and compared in patients without post-operative staple line complications vs. patients with post-operative staple line complications.
36-Item Short Form Health Survey (SF-36) | 3 weeks
  SF-36 scores will be collected at baseline and at the 3-week follow up appointment and compared for quality-of-life changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Gijos Clinic, Kaunas, Lithuania